CLINICAL TRIAL: NCT06098898
Title: Exploratory Study of NK510 Cell Therapy Combined With Monoclonal Antibody in the Treatment of Recurrent and Refractory Advanced Gastric Cancer
Brief Title: Safety and Efficacy of NK510 to Treat Gastric Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Base Therapeutics (Shanghai) Co., Ltd. (Industry)
Collaborators: Shanghai 10th People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NK510-08
Record Dates: First submitted 2023-10-17; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Intervention Model Description: Dose escalation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (low-dose NK510 monotherapy) (Experimental): NK510 9×10^9 NK cells/dose.
  Interventions: Drug: NK510
- Group B (low-dose NK510 combined mAbs) (Experimental): NK510 9×10^9 NK cells/dose. PD-1 blockade or anti-HER2 mAbs.
  Interventions: Drug: NK510; Drug: Tislelizumab，atezolizumab or Trastuzumab
- Group C (high-dose NK510 combined mAbs) (Experimental): NK510 12×10^9 NK cells/dose. PD-1 blockade or anti-HER2 mAbs.
  Interventions: Drug: NK510; Drug: Tislelizumab，atezolizumab or Trastuzumab

INTERVENTIONS:
Drug: NK510 — NK510 will be administered through intravenous infusion.3 infusions on Day 0，Day 2 and day 3 for a cycle，for a total of two cycles.
Drug: Tislelizumab，atezolizumab or Trastuzumab — Administer according to the instructions.
  Arms: Group B (low-dose NK510 combined mAbs); Group C (high-dose NK510 combined mAbs)

SUMMARY:
This study will evaluate the safety and efficacy of NK510 in the treatment of relapsed and refractory advanced gastric cancer.NK510 will be administered in combination with PD-1 blockade or monoclonal anti-HER2 antibody. Patients are required to undergo a biopsy for confirmation of tumor PD-L1 and HER2 expression and. The safety and efficacy of this treatment will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years;
* Confirmed by histology or cytology: Adenocarcinoma at the gastric or gastroesophageal junction, with locally advanced unresectable or distant metastasis. Tumor tissue can be provided for central laboratory confirmation of HER2 and PD-L1 expression status;
* Received standard treatment before screening, currently in a state of progression or recurrence of the disease;
* According to RECIST v1.1 (Solid Tumor Efficacy Evaluation Criteria), there is at least one CT measurable lesion present;
* ECOG physical status score of 0-2;
* Expected survival >=3 months;
* Except for hair loss and fatigue, all previous anti-tumor treatments have alleviated toxicity to level 1 (CTCAE v5.0) or original baseline;
* Female of childbearing age must be non lactating and have a negative serum pregnancy test within 1 week prior to enrollment;
* Able to follow the research protocol and follow-up process;
* Voluntarily sign an informed consent form to participate in this study.

Exclusion Criteria：

* Individuals who have previously discontinued treatment with trastuzumab or PD-1 monoclonal antibody due to intolerance to drug toxicity reactions;
* Pregnant or lactating female patients;
* Patients with central nervous system metastasis (CNS) and/or cancerous meningitis and obvious symptoms;
* Having other malignant tumors that require active treatment within the past 3 years;
* Subjects with active, known or suspected autoimmune diseases [excluding type I diabetes, hypothyroidism requiring hormone replacement therapy only, skin diseases not requiring systemic treatment (such as vitiligo, psoriasis or alopecia) or diseases that are not expected to recur without external triggers;
* subjects have a history of immune deficiency, including HIV testing positive, or other acquired or congenital immune deficiency diseases or organ transplantation history;
* Have a history of serious cardiovascular and cerebrovascular diseases, including but not limited to: severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, third degree atrioventricular block, etc; At rest, the QTc interval obtained from a 12 lead electrocardiogram examination is>480 ms; Acute coronary syndrome, congestive heart failure, aortic dissection,stroke, or other Grade 3 or above cardiovascular and cerebrovascular events occurred within 6 months prior to enrollment; The New York Heart Association (NYHA) has a heart function rating of ≥ II or a left ventricular ejection fraction (LVEF) of<50%; Clinically uncontrollable hypertension;
* Radical radiotherapy was performed within 4 weeks prior to enrollment;Local palliative radiotherapy or Chinese herbal medicine/traditional Chinese patent medicines and simple preparations with anti-tumor indications within 2 weeks before enrollment;
* Not fully recovered from major surgery or trauma within 2 weeks prior to enrollment;
* Participated in research drug trials and received research treatment or used research instruments within 4 weeks before enrollment;
* Other anti-tumor treatments outside of this research protocol are currently underway or planned;
* Received blood transfusion, erythropoietin, granulocyte colony stimulating factor (G-CSF), or granulocyte macrophage colony stimulating factor treatment within 2 weeks prior to enrollment;
* Subjects who received systemic treatment with corticosteroids (prednisone>10 mg/day or equivalent) or other immunosuppressive/enhancing drugs (such as thymosin, interleukin-2, and interferon) within 2 weeks prior to enrollment. Allowing selected subjects to inhale or topically use corticosteroids in the absence of active autoimmune diseases;
* The virological examination of hepatitis B or hepatitis C during screening meets any of the following criteria:

  1. HBsAg positive and peripheral blood HBV-DNA titer detection ≥ 1×10^3 copies/mL or upper limit of normal value;
  2. HCV antibody positive;
* Meet any of the following standards:

  1. Hematological:Neutrophil count <1.5×10^9/L; Platelet count <75×10^9/L; Hemoglobin < 9 g/dL;
  2. Hepatic:ALT>3×ULN (tumor liver metastasis ≥ 5×ULN); AST>3×ULN (tumor liver metastasis ≥ 5×ULN); TBIL>1.5×ULN or TBIL>2.5(3.0 mg/dL) in Gilbert syndrome subjects;
  3. Renal:Serum creatinine>1.5×ULN or creatinine clearance<50mL/min;
* Any uncertain factors that affect the safety or compliance of patients;
* Researchers believe that any other serious or uncontrollable medical disease, active infection,abnormal physical examination, laboratory examination, mental state change, or mental illness increases the risk of the subject or affects the research results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity | 6 weeks
  To evaluate the DLT during N510 treatment
Maximal Tolerable Dose | 6 weeks
  To evaluate the MTD of NK510

SECONDARY OUTCOMES:
Overall response rate (ORR) | 6 weeks
  Effectiveness Metrics

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No